CLINICAL TRIAL: NCT04134338
Title: Effect of Surgical Wound Infection on Health of Women
Brief Title: Effect of Surgical Wound Infection on Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Researcher , lecturer ,Obstetrics and Gynecology , National Research Centre, Aljazeera Hospital
Other Study IDs: surgical wound
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: To evaluate the effect of wound infection on costs — the degree of costs that is required for trating wound infection

SUMMARY:
A surgical site infection (SSI) is an infection that occurs after surgery in the part of the body

DETAILED DESCRIPTION:
Morbidity and mortality were associated with increase of surgical site infections (SSIs).Besides, it was a financial burden and negatively impact of SSIs on patient quality of life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* wound who had infection post surgery

Exclusion Criteria:

* women who had no infection

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — wound who are doing surgery
Study Population: women who experienced wound infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-10-24 (Estimated); Study Completion 2019-10-29 (Estimated)

PRIMARY OUTCOMES:
What is the effect of surgical site infection on health care cost | within a month
  how much does it cost for wound infection

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Kasralainy Hospital, Cairo, Egypt